CLINICAL TRIAL: NCT04884178
Title: Post-Market Clinical Follow-up Study of Preloaded Trifocal IOL Delivery System
Brief Title: PMCF Study of Preloaded Trifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ICARES Medicus, Inc. (Industry)
Collaborators: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPRO-000001
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Cataract
Keywords: Cataract; Trifocal; IOL; Intraocular lens; Preloaded; Aphakic; Spectacle independence; Asqelio; aspicio; AST Products; ICARES
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trifocal Preloaded IOL Delivery System (Experimental): Bilateral trifocal IOLs implanted through preloaded IOL Delivery System in the capsular bag in the posterior chamber of the eye during cataract surgery
  Interventions: Device: Trifocal Preloaded IOL Delivery System

INTERVENTIONS:
Device: Trifocal Preloaded IOL Delivery System — UV and blue-light filtering foldable trifocal IOL with a +2.2 diopter (D) addition power of intermediate visual acuity and a +3.3 D addition power of near visual acuity. This device is approved in Taiwan.
  Other Names: Asqelio Trifocal; TFPIO130Y; TFLIO130; aspicio Trifocal; PTF60Y; TF60

SUMMARY:
This is a study to evaluate the safety, effectiveness and patient satisfaction of the Trifocal Intraocular Lens after implanted to replace the natural lens following cataract removal.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of safety, effectiveness and patient satisfactions of the Trifocal Intraocular Lens after successful bilateral cataract surgery. Subjects will be assessed pre-operative, operative date and at 1-2 days, 1-2 weeks, 1-2 months, 3-4 months and 6 months post-operative. Clinical evaluations will include probability of adverse events, patient satisfaction questionnaire, as well as measurements of monocular and bilateral far, intermediate and near visual acuity as a result of Trifocal Lens performance, etc.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataracts: Adults, 20 years of age or older at the time of informed consent, of either gender, diagnosed with bilateral cataracts
* Desire for high post-operative spectacle independence
* Willingness to cooperate with and complete all post-operative visits
* Calculated lens power within +5.0 D and +34.0 D
* Planned cataract removal by phacoemulsification
* Clear intraocular media other that cataracts in both eyes
* Potential post-operative visual acuity of 20/25 or better
* Ability to comprehend and sign an informed consent
* Signed informed consent

Exclusion Criteria:

* More than 1.0 D of pre-operative corneal astigmatism
* Expected post-operative astigmatism of more than 0.75 D
* Mature/dense cataract which makes the pre-operative fundus examination difficult
* Previous ocular surgery or trauma
* Clinically significant irregular astigmatism
* Choroidal hemorrhage
* Microphthalmos
* Severe corneal dystrophy
* Medically controlled or uncontrolled glaucoma
* Clinically significant macular/RPE changes
* Concomitant severe eye disease
* Severe optic nerve atrophy
* Diabetic retinopathy, proliferative or macular edema
* Amblyopia
* Extremely shallow anterior chamber
* Chronic sever uveitis
* Pregnant or lactating
* Previous retinal detachment
* Previous corneal transplant
* Concurrent participation in another drug or device investigation
* May be expected to require other ocular surgery during the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Photopic monocular CDVA, 400 cm | 6 Months post second eye implantation
Photopic monocular CIVA, 60 cm | 6 Months post second eye implantation
Photopic monocular CNVA, 40 cm | 6 Months post second eye implantation
Rates of adverse events vs. ISO 11979-7:2018 SPE rate | 6 Months post second eye implantation

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Shiou Hwang, Dr., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan District, Taiwan